CLINICAL TRIAL: NCT00015977
Title: Phase II Study of Immunization With PSMA Peptide-Pulsed Autologous PBMC Plus rhIL-12 in Patients With Metastatic Prostate Cancer
Brief Title: Vaccine Therapy Plus Interleukin-12 in Treating Patients With Metastatic Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9845; UCCRC-9845; NCI-1192
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Interleukin-12 Subunit p35; Interleukin-12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PSMA peptide vaccine (Experimental): Immunization with PSMA peptide vaccine followed by injection of Interleukin-12 (IL-12) on Day 1 of a 21-day cycle. Additional injections of IL-12 given on Days 3 and 5 of each cycle.
  Interventions: Biological: PSA prostate cancer vaccine; Biological: recombinant interleukin-12

INTERVENTIONS:
Biological: PSA prostate cancer vaccine
Biological: recombinant interleukin-12
  Other Names: IL-12, rhIL-12

SUMMARY:
RATIONALE: Vaccines made from a patient's white blood cells may make the body build an immune response to kill cancer cells. Interleukin-12 may kill cancer cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill cancer cells. Combining vaccine therapy with interleukin-12 may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy combined with interleukin-12 in treating patients who have metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether immunization with prostate-specific membrane antigen-pulsed autologous peripheral blood mononuclear cells and interleukin-12 can promote specific T-cell priming in patients with metastatic hormone-refractory prostate cancer.
* Determine the clinical response in patients treated with this regimen.

OUTLINE: Patients receive prostate-specific membrane antigen-pulsed autologous peripheral blood mononuclear cells subcutaneously (SC) on day 1 and interleukin-12 SC on days 1, 3, and 5. Treatment repeats every 21 days for 3-9 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 37 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic adenocarcinoma of the prostate
* HLA-A2 positive
* Progressive measurable systemic disease

  * PSA at least 5 ng/mL with 2 consecutive rising PSA levels at least 1 week apart and no measurable disease OR
  * Objective evidence of disease progression by a 20% increase in the sum of longest diameter of all target lesions or evidence of new lesions by CT or bone scan regardless of PSA status
  * Lesions must be at least 1 cm to be considered measurable
  * Progressive systemic disease after discontinuation of anti-androgen therapy
* Previously treated with orchiectomy (testosterone less than 50 ng/mL) OR luteinizing hormone-releasing hormone (LHRH) analogue therapy with or without anti-androgens

  * If on LHRH analogue therapy, must continue therapy during study
* Brain metastases allowed if previously treated, clinically stable, and weaned from prior corticosteroids

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Hemoglobin greater than 9 g/dL
* Platelet count greater than 100,000/mm^3
* No active gastrointestinal bleeding

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGPT normal
* Hepatitis B surface antigen negative

Renal:

* Creatinine less than 1.5 times ULN
* Calcium less than 11 mg/dL

Cardiovascular:

* No significant cardiovascular disease
* No cardiac arrhythmia requiring therapy

Other:

* Fertile patients must use effective barrier contraception
* No intrinsic immunosuppression
* HIV negative
* No serious concurrent infection
* No psychiatric illness that would preclude study compliance
* No clinically significant autoimmune disease
* No uncontrolled peptic ulcer disease
* No history of inflammatory bowel disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy

Chemotherapy:

* Not specified

Endocrine therapy:

* See Disease Characteristics
* At least 4 weeks since prior flutamide
* At least 6 weeks since prior bicalutamide or nilutamide
* No concurrent systemic corticosteroids except physiologic replacement doses

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* No concurrent immunosuppressive drugs (e.g., cyclosporine)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2001-11; Primary Completion 2003-03 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Disease response | 63 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F. Gajewski, MD, PhD, Study Chair — University of Chicago
Locations (1):
- University of Chicago Cancer Research Center, Chicago, Illinois, United States